CLINICAL TRIAL: NCT00457834
Title: Study on the Efficacy of bi-Ventricular Pacing of Patients With Severe Heart Failure and Chronic Atrial Fibrillation
Brief Title: Bi-Ventricular Pacing in Patients With Atrial Fibrillation and Heart Failure (BIFF-Study)
Acronym: BIFF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Umeå University (Other)
Responsible Party: Steen Jensen, Heart Centre, Umeå University Hospital and Department of Public Health and Clinical Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Um dnr 03-032
Record Dates: First submitted 2007-04-04; First posted 2007-04-09 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Heart Failure
Keywords: Heart failure; Dyssynchrony; Cardiac resynchronization therapy; Atrial fibrillation; RVOT; RVapex
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

INTERVENTIONS:
Device: InSync III — Bi-ventricular pacing from leads in LV+RVA or LV+RVOT

SUMMARY:
Cardiac resynchronization therapy (CRT) is used to treat dilated heart failure with discoordinate contraction. Dyssynchrony typically stems from electrical delay leading to mechanical delay between the septal and lateral walls. Right ventricular apical pacing might be associated with long-term adverse effects on left ventricular function, and alternative pacing sites such as high septal or RVOT has been suggested. Previous studies have however been conflicting. The aim of this study is to determine if bi-ventricular pacing from RVOT + LV is better than RVapex+LV. To avoid influence from possible atrial delay only patients with chronic atrial fibrillation are included. All patients will receive a bi-ventricular pacemaker with 3 leads placed in RVapex, RVOT and via coronary sinus to pace the left ventricle. After a run in period (to determine if AV-junction ablation is necessary) the patients are randomised to one of the following pacing configurations: RVOT+LV or RVapex+LV with cross-over after 3 month.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure NYHA III-IV
* LVEF<35%
* QRS duration>150 ms
* Chronic atrial fibrillation.

Exclusion Criteria:

* Heart failure not related to systolic function
* Unstable angina pectoris, AMI, PCI or CABG within 2 month
* Inclusion in other studies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-11; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
quality of life

SECONDARY OUTCOMES:
NYHA class
6-MWT
bi-cycle test
pro-BNP
echocardiographic measures
apnea-hypopnea index

CONTACTS AND LOCATIONS:
Overall Officials: Steen M Jensen, MD, PhD, Principal Investigator — Heart Centre, Umeå University Hospital; Folke Rönn, MD, Principal Investigator — Heart Centre, Umeå University Hospital
Locations (1):
- Heart Centre, Umeå University Hospital, Umeå, Sweden

REFERENCES:
- [Derived] Ronn F, Kesek M, Karp K, Henein M, Jensen SM. Right ventricular lead positioning does not influence the benefits of cardiac resynchronization therapy in patients with heart failure and atrial fibrillation. Europace. 2011 Dec;13(12):1747-52. doi: 10.1093/europace/eur193. Epub 2011 Jun 28. PMID 21712261